CLINICAL TRIAL: NCT05886244
Title: Open-Label, Multicenter Study to Assess the Efficacy, Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Eculizumab in Complement Inhibitor Treatment Naïve Adult Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH) in China
Brief Title: Eculizumab in Adult Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH) in China
Acronym: Soliris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7414C00001
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: paroxysmal nocturnal hemoglobinuria; PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eculizumab (Experimental): Eculizumab will be administered by IV infusion.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Participants will receive 600 milligrams (mg) once a week on Day 1, 8, 15, and 22 followed by 900 mg every 2 weeks from Day 29 to Day 435.

SUMMARY:
This is a Phase 3b, single-arm, open-label, multicenter study to evaluate the efficacy, safety, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of eculizumab in adult participants with paraxysmal noturnal hemoglobinuria (PNH) in China.

DETAILED DESCRIPTION:
This is a Phase 3b, single-arm, open-label, multicenter study to evaluate the efficacy, safety, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of eculizumab in adult participants with PNH in China who previously have not been treated with complement inhibitors. Approximately 25 eligible participants in China will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adult C5 inhibitor naïve PNH patients (age>=18), which is confirmed by flow cytometry evaluation
* Must be vaccinated against N meningitidis

Exclusion Criteria:

* Meningitidis infection or unresolved meningococcal disease
* Significant bone marrow failure
* Other significant systemic diseases that might have impact on efficacy and safety assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in Lactate Dehydrogenase (LDH) at Week 12 | Baseline, Week 12
  To assess efficacy of eculizumab in participants with PNH

SECONDARY OUTCOMES:
Number(%) of participants with Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Baseline through Week 64
  To assess the safety and tolerability of eculizumab in participants with PNH
Pharmacokinetics (PK): Serum Eculizumab Concentration | Baseline through Week 64 (predose and postdose)
  To characterize the pharmacokinetics of eculizumab in participants with PNH
Change from baseline in Serum Free and total Complement 5 (C5) Concentration | Baseline through week 64 (predose and postdose)
  To characterize the pharmacodynamics of eculizumab in participants with PNH
Number(%) of participants with Antidrug Antibodies (ADAs) to Eculizumab | Baseline through Week 64
  To characterize the immunogenicity of eculizumab in participants with PNH
Change from baseline in functional assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Week 64 | Baseline through Week 64
  To assess the efficacy of eculizumab in participants with PNH
Number(%) of participants with Breakthrough Hemolysis | Baseline through Week 64
  To assess the efficacy of eculizumab in participants with PNH
Number(%) of participants achieving LDH Normalization | Baseline through Week 64
  To assess the efficacy of eculizumab in participants with PNH
Number(%) of participants needing Blood Transfusion | Baseline through Week 64
  To assess the efficacy of eculizumab in participants with PNH
Number(%) of participants changes from baseline in vital signs and laboratory parameters at all scheduled visits. | Baseline through Week 64
  To characterize the safety profile of eculizumab in participants with PNH

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Research Site, Beijing
  - Research Site, Hangzhou
  - Research Site, Nantong
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home